CLINICAL TRIAL: NCT04237896
Title: Compliance With Clinical Guidelines and Effect on Patient Outcome of Real-life Treatment of Hospitalised Exacerbations of COPD: a Nationwide Study in Spain
Brief Title: Compliance With Clinical Guidelines and Effect on Patient Outcome of Treatment of Hospitalised Exacerbations of COPD
Acronym: ADEG-EPOC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sociedad Española De Medicina Interna (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: SEMI-2019-1-COPD
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic obstructive pulmonary disease; Acute exacerbation; Inpatients; Clinical practice guidelines; Bronchodilators; Compliance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Sputum and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale. Currently there are well-established guidelines for the management of stable COPD. However, recommendations on the treatment of COPD exacerbations (E-COPD) are based on observational studies and low-quality clinical trials. In addition, there are some controversial aspects, such as treatment with systemic steroids. On the other hand, the available information on the adherence to the recommendations of the clinical practice guidelines (CPG) and its impact on the outcome of patients is scarce.

Main objectives. (1) To examine the appropriateness of two clinical guidelines (GOLD and GesEPOC) of the current management of hospitalized exacerbations of COPD; (2) To determine in real-life clinical practice the impact of adherence to CPG recommendations for management of COPD exacerbations as an outcome of the disease (stay, in-hospital mortality, and 90-days post-discharge readmissions and mortality); (3) To examine the appropriateness of two clinical guidelines (GOLD and GesEPOC) of the treatment of stable COPD at admission and after discharge in patients hospitalized with exacerbated COPD; (4) To determinate in real-life clinical practice the impact of the suitability to CPG recommendations for treatment of stable COPD on 90-day post-discharge mortality and readmission of COPD.

Method. National, multicenter, observational and longitudinal study of the first consecutive 20 patients hospitalized for exacerbations of COPD between December 10 and 23, 2019 in the Internal Medicine Services of the participating Centers. Patients will be followed 90 days after discharge. A total of 400 patients will be recruited in 20 Spanish hospitals (20 per center). Independent variables: age, sex, admission service, body mass index, dyspnea (mMRC), obstruction (FEV¬₁), exacerbations in the previous year, comorbidities, bronchodilator treatment prior to admission, criteria of adequacy to the CPG in the clinical evaluation and treatment, hyperglycemia during the first 24 hours of admission, treatment of hyperglycemia and bronchodilator treatment at discharge. Outcomes: in-hospital mortality, mortality at 90 days, re-admission at 90 days. Statistical analysis: Parametric and non-parametric tests, Kaplan-Meier and ROC curves and multiple logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Age over 40 years.
* COPD patient hospitalized with the main diagnosis of exacerbation of COPD and whose main diagnosis is confirmed by the discharge report and the local investigator.

Exclusion Criteria:

* Terminal disease
* Absence of spirometry confirmation of the COPD diagnosis.
* Presence of other diseases that can cause symptoms like those of a COPD exacerbation (e.g. heart failure, pneumonia, etc.), where exacerbation of COPD is not the main cause of admission.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 40 years who have required a hospital stay for an exacerbation of COPD prospectively followed 90 days after discharge.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-27 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
IN-HOSPITAL MORTALITY | during the admission of the index episode
  death from any cause
30-day MORTALITY | <30 days
  death from any cause
90-day MORTALITY | 31-90 days
  death from any cause
30-day READMISSIONS | < 30 days
  Readmission for an exacerbation of COPD
30-day READMISSIONS | 31-90 days
  Readmission for an exacerbation of COPD

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Medrano, Principal Investigator — Sociedad Española De Medicina Interna
Locations (1):
- Virgen del Rocío University Hospital, Seville, Spain/Seville, Spain

IPD SHARING:
Plan to Share IPD: No